CLINICAL TRIAL: NCT01803074
Title: Randomized, Placebo-Controlled, Multiple-Dose Study to Evaluate the Pharmacodynamics, Safety and Pharmacokinetics of BMS-955176 (Double-Blinded) and BMS-955176 With Atazanavir +/- Ritonavir (Open-Labeled) in HIV-1 Infected Subjects
Brief Title: Study to Evaluate a HIV Drug for the Treatment of HIV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 206739; 2012-004124-38 (EudraCT Number); AI468-002 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2013-03-01; First posted 2013-03-04 (Estimated); Results first posted 2019-11-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Infection, Human Immunodeficiency Virus; HIV Infections
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; HIV Infections | interventions — BMS-955176; Atazanavir Sulfate; Ritonavir; Tenofovir; Emtricitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (13):
- Part A-Group 1: BMS-955176 (5 mg) or Placebo (Experimental): BMS-955176 5 mg solution by mouth once daily for 10 days
  OR
  Placebo matching with BMS-955176 0 mg solution by mouth once daily for 10 days
  Interventions: Drug: BMS-955176; Drug: Placebo matching with BMS-955176
- Part A-Group 2: BMS-955176 (10 mg) or Placebo (Experimental): BMS-955176 10 mg solution by mouth once daily for 10 days
  OR
  Placebo matching with BMS-955176 0 mg solution by mouth once daily for 10 days
  Interventions: Drug: BMS-955176; Drug: Placebo matching with BMS-955176
- Part A-Group 3: BMS-955176 (20 mg) or Placebo (Experimental): BMS-955176 20 mg solution by mouth once daily for 10 days
  OR
  Placebo matching with BMS-955176 0 mg solution by mouth once daily for 10 days
  Interventions: Drug: BMS-955176; Drug: Placebo matching with BMS-955176
- Part A-Group 4: BMS-955176 (40 mg) or Placebo (Experimental): BMS-955176 40 mg solution by mouth once daily for 10 days
  OR
  Placebo matching with BMS-955176 0 mg solution by mouth once daily for 10 days
  Interventions: Drug: BMS-955176; Drug: Placebo matching with BMS-955176
- Part B-Group 5: BMS-955176 + Atazanavir (Experimental): BMS-955176 40 mg solution by mouth once daily for 28 days
  Atazanavir 2 x 200 mg capsules by mouth once daily for 28 days
  Interventions: Drug: BMS-955176; Drug: Atazanavir
- Part B-Group 6: BMS-955176 + Atazanavir + Ritonavir (Experimental): BMS-955176 40 mg solution by mouth once daily for 28 days
  Atazanavir 1 x 300 mg capsules by mouth once daily for 28 days
  Ritonavir 1 x 100 mg tablet by mouth once daily for 28 days
  Interventions: Drug: BMS-955176; Drug: Atazanavir; Drug: Ritonavir
- Part B-Group 7: Atazanavir+Ritonavir+Tenofovir+Emtricitabine (Experimental): Atazanavir 1 x 300 mg capsule by mouth once daily for 28 days
  Ritonavir 1 x 100 mg tablet by mouth once daily for 28 days
  Tenofovir 1 x 300 mg tablet by mouth once daily for 28 days
  Emtricitabine 1 x 200 mg capsule once daily for 28 days
  Interventions: Drug: Atazanavir; Drug: Ritonavir; Drug: Tenofovir; Drug: Emtricitabine
- Part C-Group 8: BMS-955176 (40 mg) or Placebo (Experimental): BMS-955176 40 mg solution by mouth once daily for 10 days
  OR
  Placebo matching with BMS-955176 0 mg solution by mouth once daily for 10 days
  Interventions: Drug: BMS-955176; Drug: Placebo matching with BMS-955176
- Part A-Group 9: BMS-955176 (80 mg) or Placebo (Experimental): BMS-955176 80 mg solution by mouth once daily for 10 days
  OR
  Placebo matching with BMS-955176 0 mg solution by mouth once daily for 10 days
  Interventions: Drug: BMS-955176; Drug: Placebo matching with BMS-955176
- Part A-Group 10: BMS-955176 (120 mg) or Placebo (Experimental): BMS-955176 120 mg solution by mouth once daily for 10 days
  OR
  Placebo matching with BMS-955176 0 mg solution by mouth once daily for 10 days
  Interventions: Drug: BMS-955176; Drug: Placebo matching with BMS-955176
- Part A-Group 11 (Optional): BMS-955176 (≤120 mg) or Placebo (Experimental): BMS-955176 ≤120 mg solution by mouth once daily for 14 days
  OR
  Placebo matching with BMS-955176 0 mg solution by mouth once daily for 14 days
  Interventions: Drug: BMS-955176; Drug: Placebo matching with BMS-955176
- Part B-Group 12: BMS-955176 (80 mg) + Atazanavir (Experimental): BMS-955176 80 mg solution by mouth once daily for 28 days
  Atazanavir 2 x 200 mg capsules by mouth once daily for 28 days
  Interventions: Drug: BMS-955176; Drug: Atazanavir
- Part C-Group 13: BMS-955176 (120 mg) or Placebo (Experimental): BMS-955176 120 mg solution by mouth once daily for 10 days
  OR
  Placebo matching with BMS-955176 0 mg solution by mouth once daily for 10 days
  Interventions: Drug: BMS-955176; Drug: Placebo matching with BMS-955176

INTERVENTIONS:
Drug: BMS-955176 — BMS-955176
  Arms: Part A-Group 10: BMS-955176 (120 mg) or Placebo; Part A-Group 11 (Optional): BMS-955176 (≤120 mg) or Placebo; Part A-Group 1: BMS-955176 (5 mg) or Placebo; Part A-Group 2: BMS-955176 (10 mg) or Placebo; Part A-Group 3: BMS-955176 (20 mg) or Placebo; Part A-Group 4: BMS-955176 (40 mg) or Placebo; Part A-Group 9: BMS-955176 (80 mg) or Placebo; Part B-Group 12: BMS-955176 (80 mg) + Atazanavir; Part B-Group 5: BMS-955176 + Atazanavir; Part B-Group 6: BMS-955176 + Atazanavir + Ritonavir; Part C-Group 13: BMS-955176 (120 mg) or Placebo; Part C-Group 8: BMS-955176 (40 mg) or Placebo
Drug: Placebo matching with BMS-955176 — Placebo matching with BMS-955176
  Arms: Part A-Group 10: BMS-955176 (120 mg) or Placebo; Part A-Group 11 (Optional): BMS-955176 (≤120 mg) or Placebo; Part A-Group 1: BMS-955176 (5 mg) or Placebo; Part A-Group 2: BMS-955176 (10 mg) or Placebo; Part A-Group 3: BMS-955176 (20 mg) or Placebo; Part A-Group 4: BMS-955176 (40 mg) or Placebo; Part A-Group 9: BMS-955176 (80 mg) or Placebo; Part C-Group 13: BMS-955176 (120 mg) or Placebo; Part C-Group 8: BMS-955176 (40 mg) or Placebo
Drug: Atazanavir — Atazanavir
  Arms: Part B-Group 12: BMS-955176 (80 mg) + Atazanavir; Part B-Group 5: BMS-955176 + Atazanavir; Part B-Group 6: BMS-955176 + Atazanavir + Ritonavir; Part B-Group 7: Atazanavir+Ritonavir+Tenofovir+Emtricitabine
Drug: Ritonavir — Ritonavir
  Arms: Part B-Group 6: BMS-955176 + Atazanavir + Ritonavir; Part B-Group 7: Atazanavir+Ritonavir+Tenofovir+Emtricitabine
Drug: Tenofovir — Tenofovir
  Arms: Part B-Group 7: Atazanavir+Ritonavir+Tenofovir+Emtricitabine
Drug: Emtricitabine — Emtricitabine
  Arms: Part B-Group 7: Atazanavir+Ritonavir+Tenofovir+Emtricitabine

SUMMARY:
The primary purpose of this study is to study the safety and tolerability of a HIV drug and to evaluate a decrease of HIV-1 virus level in blood after treatments in HIV-1 infected patients

DETAILED DESCRIPTION:
Masking: Open-Part B. Double Blind-Parts A and C

Gender: Both female and male participants for Parts A and C. Male participants for Part B.

HIV = Human Immunodeficiency Virus RNA = Ribonucleic acid

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Age 18-55 years inclusive
* Men and women: (Parts A and C); men only (Part B)
* Women of childbearing potential (WOCBP) must not be pregnant and nursing
* BMI: 18.0-35.0 kg/m2
* Subjects are infected with HIV-1 (clades B or C) and meet following criteria at the screening:

  i) Plasma HIV-1 RNA ≥5,000 copies/mL; ii) Antiretroviral treatment naive (defined as <1 week of ARV treatment) or ART-experienced (protease inhibitor and/or maturation inhibitor naive); iii) Subjects are not eligible for HIV-1 treatment based on the United States Department of Health and Human Services Panel on Antiretroviral Guidelines for Adults and Adolescents or have declined initiation of cART iv) CD4+ lymphocyte measurement ≥200 cells/μL; v) In Parts A and B, all subjects are infected with HIV-1 clade B vi) In Part C, all subjects are infected with HIV-1 clade C

Exclusion Criteria:

* History of genotypic and/or phenotypic drug resistance testing showing resistance to protease inhibitors
* Any significant acute or chronic medical illness which is not stable or is not controlled with medication or not consistent with HIV-1 infection
* Receive antiretroviral treatment within 12 weeks prior to screening
* Currently co-infected with hepatitis C or hepatitis B
* Previously received an HIV maturation inhibitor or HIV protease inhibitor
* Current or recent (within 3 months of study drug administration) gastrointestinal disease
* Any major surgery within 4 weeks of study drug administration
* Acute diarrhea lasting ≥1 day, within 3 weeks prior to randomization
* Subjects with history of Gilbert's syndrome
* Subjects previously received an HIV maturation inhibitor or HIV protease inhibitor
* A personal history of clinically relevant cardiac disease, symptomatic or asymptomatic arrhythmias, syncopal episodes, or additional risk factors for torsades de pointes. A personal or family history of long QT syndrome
* Patients who are unwilling to practice adequate infection protection during and after study participation to minimize potential for spread of HIV infection, including HIV which may have developed resistance to HIV maturation inhibitor and/or ATV
* Any gastrointestinal surgery that could impact upon the absorption of study drug
* Smoking >10 cigarettes per day
* PR ≥210 msec; QRS ≥120 msec; QT ≥500 msec; and QTcF ≥470 msec for women and ≥450 msec for men
* Evidence of second or third degree heart block prior to study drug
* Absolute Neutrophil Count <(ANC) 0.7 x lower limit of normal (LLN)
* Hemoglobin <0.8 x LLN
* Alanine aminotransferase (ALT) >1.25 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) >1.25 x ULN
* Total Bilirubin >1.25 x ULN
* Creatinine clearance <60 mL/mim
* Positive urine screen for drugs of abuse without a valid prescription (subjects positive for cannabinoids and/or amphetamines will be included)
* Positive blood screen for hepatitis C virus (HCV) RNA, hepatitis B surface antigen (consistent with active or chronic hepatitis B), or HIV-2 antibody
* History of any significant drug allergy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2013-04-04 (Actual); Primary Completion 2014-11-29 (Actual); Study Completion 2014-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Berlin, Germany

REFERENCES:
- [Derived] Hwang C, Schurmann D, Sobotha C, Boffito M, Sevinsky H, Ray N, Ravindran P, Xiao H, Keicher C, Huser A, Krystal M, Dicker IB, Grasela D, Lataillade M. Antiviral Activity, Safety, and Exposure-Response Relationships of GSK3532795, a Second-Generation Human Immunodeficiency Virus Type 1 Maturation Inhibitor, Administered as Monotherapy or in Combination With Atazanavir With or Without Ritonavir in a Phase 2a Randomized, Dose-Ranging, Controlled Trial (AI468002). Clin Infect Dis. 2017 Aug 1;65(3):442-452. doi: 10.1093/cid/cix239. PMID 28369211
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 3 centers in 3 countries (1 in Germany, 1 in the United Kingdom, 1 in South Africa) from 04-April-2013 to 29-November-2014.
Pre-assignment Details: Participants screened were 191 of which 84 were screen failures (Participant withdrew consent: 3, Pregnancy: 3, Participant no longer meets study criteria: 73, Not according to participant's schedule: 1, Not included since cohort was closed: 3 and back up participant: 1). Only 107 participants (Part A: 60; Part B: 28; and Part C: 19) were enrolled.
Groups:
- Part A-Group 1: BMS-955176 (5 mg): Participants infected with Human Immunodeficiency Virus Type-1 (HIV-1) clade B were treated with 5 milligrams (mg) BMS-955176 as oral suspension, once daily (QD) from Day 1 to Day 10. Participants were evaluated for a total period of 24 days from the day of first dose.
- Part A-Group 2: BMS-955176 (10 mg): Participants infected with HIV-1 clade B were treated with 10 mg BMS-955176 as oral suspension, QD from Day 1 to Day 10. Participants were evaluated for a total period of 24 days from the day of first dose.
- Part A-Group 3: BMS-955176 (20 mg): Participants infected with HIV-1 clade B were treated with 20 mg BMS-955176 as oral suspension, QD from Day 1 to Day 10. Participants were evaluated for a total period of 24 days from the day of first dose.
- Part A-Group 4: BMS-955176 (40 mg): Participants infected with HIV-1 clade B were treated with 40 mg BMS-955176 as oral suspension, QD from Day 1 to Day 10. Participants were evaluated for a total period of 24 days from the day of first dose.
- Part A-Group 9: BMS-955176 (80 mg): Participants infected with HIV-1 clade B were treated with 80 mg BMS-955176 as oral suspension, QD from Day 1 to Day 10 under fasting condition. Participants were evaluated for a total period of 24 days from the day of first dose.
- Part A-Group 10: BMS-955176 (120 mg): Participants infected with HIV-1 clade B were treated with 120 mg BMS-955176 as oral suspension, QD from Day 1 to Day 10 under fasting condition. Participants were evaluated for a total period of 24 days from the day of first dose.
- Placebo Clade B: Participants infected with HIV-1 clade B were treated with matching placebo QD from Day 1 to Day 10. Participants were evaluated for a total period of 24 days from the day of first dose.
- Part B-Group 5: BMS-955176 (40 mg) + Atazanavir: Participants infected with HIV-1 clade B were treated with 40 mg BMS 955176 as oral suspension and 400 mg atazanavir (2*200 mg) capsules, QD from Day 1 to Day 28 with breakfast. Participants were evaluated for a total period of 42 days from the day of first dose.
- Part B-Group 6: BMS-955176 (40 mg) + Atazanavir + Ritonavir: Participants infected with HIV-1 clade B were treated with 40 mg BMS-955176 as oral suspension, 300 mg atazanavir capsules and 100 mg ritonavir tablets, QD from Day 1 to Day 28 with breakfast. Participants were evaluated for a total period of 42 days from the day of first dose.
- Part B-Group 7: Atazanavir+Ritonavir+Tenofovir+Emtricitabine: Participants infected with HIV-1 clade B were treated with 300 mg tenofovir, 200 mg emtricitabine, 300 mg atazanavir capsules and 100 mg ritonavir tablets, QD from Day 1 to Day 28 with breakfast. Participants were evaluated for a total period of 42 days from the day of first dose.
- Part B-Group 12: BMS-955176 (80 mg) + Atazanavir: Participants infected with HIV-1 clade B were treated with 80 mg BMS-955176 as oral suspension and 400 mg atazanavir (2*200 mg) capsules, QD from Day 1 to Day 28 with breakfast. Participants were evaluated for a total period of 42 days from the day of first dose.
- Part C-Group 8: BMS-955176 (40 mg): Participants infected with HIV-1 clade C were treated with 40 mg BMS-955176 as oral suspension, QD from Day 1 to Day 10. Participants were evaluated for a total period of 24 days from the day of first dose.
- Part C-Group 13: BMS-955176 (120 mg): Participants infected with HIV-1 clade C were treated with 120 mg BMS-955176 as oral suspension, QD from Day 1 to Day 10. Participants were evaluated for a total period of 24 days from the day of first dose.
- Placebo Clade C: Participants infected with HIV-1 clade C were treated with matching placebo, QD from Day 1 to Day 10. Participants were evaluated for a total period of 24 days from the day of first dose.
Period: Period 1: Part A (HIV-1 Clade B)
Arm/Group | Part A-Group 1: BMS-955176 (5 mg) | Part A-Group 2: BMS-955176 (10 mg) | Part A-Group 3: BMS-955176 (20 mg) | Part A-Group 4: BMS-955176 (40 mg) | Part A-Group 9: BMS-955176 (80 mg) | Part A-Group 10: BMS-955176 (120 mg) | Placebo Clade B | Part B-Group 5: BMS-955176 (40 mg) + Atazanavir | Part B-Group 6: BMS-955176 (40 mg) + Atazanavir + Ritonavir | Part B-Group 7: Atazanavir+Ritonavir+Tenofovir+Emtricitabine | Part B-Group 12: BMS-955176 (80 mg) + Atazanavir | Part C-Group 8: BMS-955176 (40 mg) | Part C-Group 13: BMS-955176 (120 mg) | Placebo Clade C
Started | 8 | 8 | 8 | 8 | 8 | 8 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 8 | 8 | 8 | 8 | 8 | 8 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2: Part B (HIV-1 Clade B)
Arm/Group | Part A-Group 1: BMS-955176 (5 mg) | Part A-Group 2: BMS-955176 (10 mg) | Part A-Group 3: BMS-955176 (20 mg) | Part A-Group 4: BMS-955176 (40 mg) | Part A-Group 9: BMS-955176 (80 mg) | Part A-Group 10: BMS-955176 (120 mg) | Placebo Clade B | Part B-Group 5: BMS-955176 (40 mg) + Atazanavir | Part B-Group 6: BMS-955176 (40 mg) + Atazanavir + Ritonavir | Part B-Group 7: Atazanavir+Ritonavir+Tenofovir+Emtricitabine | Part B-Group 12: BMS-955176 (80 mg) + Atazanavir | Part C-Group 8: BMS-955176 (40 mg) | Part C-Group 13: BMS-955176 (120 mg) | Placebo Clade C
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 4 | 8 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 4 | 8 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3: Part C (HIV-1 Clade C Only)
Arm/Group | Part A-Group 1: BMS-955176 (5 mg) | Part A-Group 2: BMS-955176 (10 mg) | Part A-Group 3: BMS-955176 (20 mg) | Part A-Group 4: BMS-955176 (40 mg) | Part A-Group 9: BMS-955176 (80 mg) | Part A-Group 10: BMS-955176 (120 mg) | Placebo Clade B | Part B-Group 5: BMS-955176 (40 mg) + Atazanavir | Part B-Group 6: BMS-955176 (40 mg) + Atazanavir + Ritonavir | Part B-Group 7: Atazanavir+Ritonavir+Tenofovir+Emtricitabine | Part B-Group 12: BMS-955176 (80 mg) + Atazanavir | Part C-Group 8: BMS-955176 (40 mg) | Part C-Group 13: BMS-955176 (120 mg) | Placebo Clade C
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 7 | 4
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 7 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part A-Group 1: BMS-955176 (5 mg): Participants infected with HIV-1 clade B were treated with 5 mg BMS-955176 as oral suspension, QD from Day 1 to Day 10. Participants were evaluated for a total period of 24 days from the day of first dose.
- Total: Total of all reporting groups
Arm/Group | Part A-Group 1: BMS-955176 (5 mg) | Part A-Group 2: BMS-955176 (10 mg) | Part A-Group 3: BMS-955176 (20 mg) | Part A-Group 4: BMS-955176 (40 mg) | Part A-Group 9: BMS-955176 (80 mg) | Part A-Group 10: BMS-955176 (120 mg) | Placebo Clade B | Part B-Group 5: BMS-955176 (40 mg) + Atazanavir | Part B-Group 6: BMS-955176 (40 mg) + Atazanavir + Ritonavir | Part B-Group 7: Atazanavir+Ritonavir+Tenofovir+Emtricitabine | Part B-Group 12: BMS-955176 (80 mg) + Atazanavir | Part C-Group 8: BMS-955176 (40 mg) | Part C-Group 13: BMS-955176 (120 mg) | Placebo Clade C | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 12 | 8 | 8 | 4 | 8 | 8 | 7 | 4 | 107
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.6 (8.73) | 37.5 (11.07) | 33.3 (7.19) | 39.5 (8.09) | 36.3 (11.23) | 38.0 (9.49) | 36.3 (7.12) | 33.0 (7.21) | 36.3 (9.24) | 32.8 (10.21) | 34.3 (6.80) | 33.6 (7.80) | 35.4 (9.59) | 35.3 (8.54) | 36.1 (8.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 8
  Male | 8 | 7 | 8 | 8 | 8 | 8 | 12 | 8 | 8 | 4 | 8 | 5 | 5 | 2 | 99
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 7 | 8 | 8 | 8 | 8 | 12 | 6 | 8 | 4 | 7 | 2 | 0 | 0 | 84
  Black/African American | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 7 | 3 | 17
  American Indian/Alaska | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Other | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Plasma Log10 HIV-1 Ribonucleic Acid (RNA) Levels From Baseline to Day 11
Description: Antiviral activity of BMS-955176 was estimated by measuring the plasma HIV-1 RNA levels in the HIV-1 infected participants. Change in the plasma HIV-1 RNA levels were measured in the participants infected with HIV-1 clade B and C who received BMS-955176 monotherapy. Baseline was Day 1. Change from Baseline was post-Baseline individual values minus Baseline values.
Time Frame: Baseline (Day 1) and Day 11 after the final dose with BMS-955176
Population: All Treated Subjects Population comprised of all participants who had received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Log10 copies per milliliter (c/mL)
Arm/Group | Part A-Group 1: BMS-955176 (5 mg) | Part A-Group 2: BMS-955176 (10 mg) | Part A-Group 3: BMS-955176 (20 mg) | Part A-Group 4: BMS-955176 (40 mg) | Part A-Group 9: BMS-955176 (80 mg) | Part A-Group 10: BMS-955176 (120 mg) | Part B-Group 5: BMS-955176 (40 mg) + Atazanavir | Part B-Group 6: BMS-955176 (40 mg) + Atazanavir + Ritonavir | Part B-Group 7: Atazanavir+Ritonavir+Tenofovir+Emtricitabine | Part B-Group 12: BMS-955176 (80 mg) + Atazanavir | Part C-Group 8: BMS-955176 (40 mg) | Part C-Group 13: BMS-955176 (120 mg) | Placebo Clade B | Placebo Clade C
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 4 | 8 | 8 | 7 | 12 | 4
Log10 copies per milliliter (c/mL) | -0.138 (0.1281) | -0.567 (0.5845) | -0.889 (0.6582) | -1.279 (0.4596) | -1.339 (0.29) | -1.326 (0.3855) | -1.216 (0.4366) | -1.431 (0.2967) | -1.544 (0.4155) | -1.521 (0.2651) | -1.29 (0.3376) | -0.938 (0.6897) | 0.118 (0.5277) | -0.172 (0.7876)

2. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) - Part A and C
Description: Time to reach the maximum plasma concentration was directly determined from concentration time data.
Time Frame: Pre-dose Day 1 and Day 10
Population: Pharmacokinetic Population comprised of all participants who received any study medication and had any available concentration-time data.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A-Group 1: BMS-955176 (5 mg) | Part A-Group 2: BMS-955176 (10 mg) | Part A-Group 3: BMS-955176 (20 mg) | Part A-Group 4: BMS-955176 (40 mg) | Part A-Group 9: BMS-955176 (80 mg) | Part A-Group 10: BMS-955176 (120 mg) | Part C-Group 8: BMS-955176 (40 mg) | Part C-Group 13: BMS-955176 (120 mg)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 7
Hours
  Day 1 | 3 [1.5 to 6] | 2.51 [2 to 4] | 3 [3 to 6] | 4 [2 to 6] | 3.5 [3 to 4] | 3 [1.5 to 6] | 3.5 [2 to 10] | 3.53 [2 to 4.25]
  Day 10 | 3 [2 to 4] | 3 [1.5 to 4] | 4 [3 to 16] | 3 [2 to 6] | 3 [1.5 to 4.02] | 2.5 [1.5 to 3.87] | 3 [2 to 6] | 3 [1.55 to 4]

3. Secondary Outcome: Number of Participants With Death as Outcome, Serious Adverse Events (SAEs), Related SAEs, Discontinuations Due to SAEs, Adverse Events (AEs), and Discontinuations Due to AEs During the Study
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Related=having certain, probable, possible, or unknown relationship to study drug.
Time Frame: Day 1 to end of the study (Day 42)
Population: All Treated Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-Group 1: BMS-955176 (5 mg) | Part A-Group 2: BMS-955176 (10 mg) | Part A-Group 3: BMS-955176 (20 mg) | Part A-Group 4: BMS-955176 (40 mg) | Part A-Group 9: BMS-955176 (80 mg) | Part A-Group 10: BMS-955176 (120 mg) | Part B-Group 5: BMS-955176 (40 mg) + Atazanavir | Part B-Group 6: BMS-955176 (40 mg) + Atazanavir + Ritonavir | Part B-Group 7: Atazanavir+Ritonavir+Tenofovir+Emtricitabine | Part B-Group 12: BMS-955176 (80 mg) + Atazanavir | Part C-Group 8: BMS-955176 (40 mg) | Part C-Group 13: BMS-955176 (120 mg) | Placebo Clade B | Placebo Clade C
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 4 | 8 | 8 | 7 | 12 | 4
Participants
  Deaths | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Discontinuations due to SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Discontinuations due to AEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AEs | 5 | 5 | 5 | 6 | 8 | 7 | 8 | 8 | 4 | 6 | 7 | 6 | 9 | 3

4. Secondary Outcome: Maximum Decline From Baseline in Log10 HIV-1 RNA - Part A and C
Description: Antiviral activity of BMS-955176 was estimated by measuring the plasma HIV-1 RNA levels in the HIV-1 infected participants. Maximum decline from Baseline in the plasma HIV-1 RNA levels were measured in the participants infected with HIV-1 clade B and C. Baseline was Day 1. Change from Baseline was post-Baseline individual values minus Baseline values.
Time Frame: Baseline (Day 1) up to Day 24
Population: All Treated Subjects Population.
Measure: Median (Full Range); unit: Log10 copies/mL
Arm/Group | Part A-Group 1: BMS-955176 (5 mg) | Part A-Group 2: BMS-955176 (10 mg) | Part A-Group 3: BMS-955176 (20 mg) | Part A-Group 4: BMS-955176 (40 mg) | Part A-Group 9: BMS-955176 (80 mg) | Part A-Group 10: BMS-955176 (120 mg) | Part C-Group 8: BMS-955176 (40 mg) | Part C-Group 13: BMS-955176 (120 mg) | Placebo Clade B | Placebo Clade C
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 7 | 12 | 4
Log10 copies/mL | -0.498 [-0.78 to -0.22] | -0.976 [-1.76 to -0.64] | -1.115 [-2.12 to -0.13] | -1.701 [-1.88 to -0.93] | -1.555 [-1.82 to -1.04] | -1.654 [-2.07 to -0.83] | -1.352 [-2.03 to -1.04] | -1.257 [-2.02 to -0.7] | -0.381 [-1.46 to 0.56] | -0.419 [-1.21 to 0.22]

5. Secondary Outcome: Maximum Decline From Baseline in Log10 HIV-1 RNA - Part B
Description: as for outcome 4
Time Frame: Baseline (Day 1) up to Day 42
Population: All Treated Subjects Population.
Measure: Median (Full Range); unit: Log10 copies/mL
Arm/Group | Part B-Group 5: BMS-955176 (40 mg) + Atazanavir | Part B-Group 6: BMS-955176 (40 mg) + Atazanavir + Ritonavir | Part B-Group 7: Atazanavir+Ritonavir+Tenofovir+Emtricitabine | Part B-Group 12: BMS-955176 (80 mg) + Atazanavir
Number analyzed (Participants) | 8 | 8 | 4 | 8
Log10 copies/mL | -1.858 [-2.37 to -1.49] | -2.202 [-3.52 to -1.24] | -2.39 [-3.04 to -1.83] | -2.228 [-2.68 to -1.87]

6. Secondary Outcome: Time to Maximum Decline in Log 10 HIV-1 RNA - Part A and C
Description: Antiviral activity of BMS-955176 was estimated by measuring the plasma HIV-1 RNA levels in the HIV-1 infected participants. Time to maximum decline in the plasma HIV-1 RNA levels were measured in the participants infected with HIV-1 clade B and C. Baseline was Day 1. Change from Baseline was post-Baseline individual values minus Baseline values.
Time Frame: Baseline (Day 1) up to Day 24
Population: All Treated Subjects Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A-Group 1: BMS-955176 (5 mg) | Part A-Group 2: BMS-955176 (10 mg) | Part A-Group 3: BMS-955176 (20 mg) | Part A-Group 4: BMS-955176 (40 mg) | Part A-Group 9: BMS-955176 (80 mg) | Part A-Group 10: BMS-955176 (120 mg) | Part C-Group 8: BMS-955176 (40 mg) | Part C-Group 13: BMS-955176 (120 mg) | Placebo Clade B | Placebo Clade C
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 7 | 12 | 4
Hours | 168 [72 to 433.4] | 216 [48 to 553.5] | 203.9 [168 to 288.1] | 240.15 [120.1 to 312.1] | 204 [168 to 384.6] | 240.2 [216 to 288.3] | 228.05 [192 to 384.6] | 215.8 [120 to 312] | 216.2 [24 to 433.8] | 132.05 [23.9 to 786.3]

7. Secondary Outcome: Time to Maximum Decline in Log 10 HIV-1 RNA - Part B
Description: as for outcome 6
Time Frame: Baseline (Day 1) up to Day 42
Population: All Treated Subjects Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part B-Group 5: BMS-955176 (40 mg) + Atazanavir | Part B-Group 6: BMS-955176 (40 mg) + Atazanavir + Ritonavir | Part B-Group 7: Atazanavir+Ritonavir+Tenofovir+Emtricitabine | Part B-Group 12: BMS-955176 (80 mg) + Atazanavir
Number analyzed (Participants) | 8 | 8 | 4 | 8
Hours | 624 [360 to 816] | 636.05 [216 to 816.9] | 588 [528 to 672.1] | 636.05 [528 to 816.3]

8. Secondary Outcome: Change From Baseline in Cluster of Differentiation (CD) 4+ and CD8+ Lymphocyte Counts - Part A and C
Description: Change in the CD4+ and CD8+ cell counts from Baseline were measured in the participants infected with HIV-1 clade B and C who received BMS-955176 + ATV or BMS-955176 + ATV + RTV therapy. Baseline was Day 1. Change from Baseline was post-Baseline individual values minus Baseline values.
Time Frame: Baseline (Day 1) up to Day 24
Population: All Treated Subjects Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Cells/microliter
Arm/Group | Part A-Group 1: BMS-955176 (5 mg) | Part A-Group 2: BMS-955176 (10 mg) | Part A-Group 3: BMS-955176 (20 mg) | Part A-Group 4: BMS-955176 (40 mg) | Part A-Group 9: BMS-955176 (80 mg) | Part A-Group 10: BMS-955176 (120 mg) | Part C-Group 8: BMS-955176 (40 mg) | Part C-Group 13: BMS-955176 (120 mg) | Placebo Clade B | Placebo Clade C
Number analyzed (Participants) | 6 | 7 | 7 | 7 | 8 | 7 | 6 | 6 | 9 | 4
Cells/microliter
  CD4+ | -21.8 (88.37) | 14.6 (120.82) | -70.1 (68.49) | -23.6 (42.13) | -43.8 (69.5) | -56.7 (78.26) | -53.7 (93.76) | 24.5 (57.58) | -77.3 (91.05) | 18 (67.3)
  CD8+ | -95 (301.52) | -8.3 (236.48) | -107.4 (264.26) | -57.3 (126.25) | -194.6 (182.3) | -161.3 (203.01) | -214.4 (390.13) | -155.8 (56.55) | -93.1 (138.52) | -136.3 (224.49)

9. Secondary Outcome: Change From Baseline in Cluster of Differentiation (CD) 4+ and CD8+ Lymphocyte Counts - Part B
Description: as for outcome 8
Time Frame: Baseline (Day 1) up to Day 42
Population: All Treated Subjects Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Cells/microliter
Arm/Group | Part B-Group 5: BMS-955176 (40 mg) + Atazanavir | Part B-Group 6: BMS-955176 (40 mg) + Atazanavir + Ritonavir | Part B-Group 7: Atazanavir+Ritonavir+Tenofovir+Emtricitabine | Part B-Group 12: BMS-955176 (80 mg) + Atazanavir
Number analyzed (Participants) | 5 | 7 | 4 | 4
Cells/microliter
  CD4+ | -133.2 (84.14) | -106.4 (166.59) | 33 (144.79) | -89 (35.71)
  CD8+ | -442.8 (243.99) | -466.1 (491.21) | -216.3 (287.06) | -147 (140.67)

10. Secondary Outcome: Percent Change From Baseline in Cluster of Differentiation (CD) 4+ and CD8+ Lymphocyte Percent - Part A and C
Description: Percent Change in the CD4+ and CD8+ cell counts from Baseline were measured in the participants infected with HIV-1 clade B and C who received BMS-955176 + ATV or BMS-955176 + ATV + RTV therapy. Baseline was Day 1. Change from Baseline was post-Baseline individual values minus Baseline values.
Time Frame: Baseline (Day 1) up to Day 24
Population: All Treated Subjects Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Part A-Group 1: BMS-955176 (5 mg) | Part A-Group 2: BMS-955176 (10 mg) | Part A-Group 3: BMS-955176 (20 mg) | Part A-Group 4: BMS-955176 (40 mg) | Part A-Group 9: BMS-955176 (80 mg) | Part A-Group 10: BMS-955176 (120 mg) | Part C-Group 8: BMS-955176 (40 mg) | Part C-Group 13: BMS-955176 (120 mg) | Placebo Clade B | Placebo Clade C
Number analyzed (Participants) | 6 | 7 | 7 | 7 | 8 | 7 | 6 | 6 | 9 | 4
Percent change
  CD4+ | 2.33 (2.944) | 0.29 (2.215) | -1.29 (5.057) | 0.86 (3.288) | 2.13 (3.399) | 0.29 (2.87) | 0.5 (3.017) | 3.17 (3.371) | -0.22 (3.93) | 2.75 (3.775)
  CD8+ | 1.17 (2.401) | 0.43 (3.207) | 0 (6.325) | 1 (3.225) | -0.25 (5.064) | -2.29 (2.812) | 0 (1.871) | -4.25 (3.775) | 1.75 (4.2) | -1.33 (5.132)

11. Secondary Outcome: Percent Change From Baseline in Cluster of Differentiation (CD) 4+ and CD8+ Lymphocyte Percent - Part B
Description: as for outcome 10
Time Frame: Baseline (Day 1) up to Day 42
Population: All Treated Subjects Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Part B-Group 5: BMS-955176 (40 mg) + Atazanavir | Part B-Group 6: BMS-955176 (40 mg) + Atazanavir + Ritonavir | Part B-Group 7: Atazanavir+Ritonavir+Tenofovir+Emtricitabine | Part B-Group 12: BMS-955176 (80 mg) + Atazanavir
Number analyzed (Participants) | 5 | 8 | 4 | 4
Percent change
  CD4+ | 2.4 (2.881) | 3.25 (3.105) | 4.75 (2.217) | -0.75 (1.893)
  CD8+ | -2.8 (1.924) | -6.25 (4.464) | -3.75 (2.062) | -1.25 (2.217)

12. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) - Part B
Description: Tmax was directly determined from concentration time data.
Time Frame: Pre-dose Day 1 and Day 28
Population: Pharmacokinetic Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part B-Group 5: BMS-955176 (40 mg) + Atazanavir | Part B-Group 6: BMS-955176 (40 mg) + Atazanavir + Ritonavir | Part B-Group 12: BMS-955176 (80 mg) + Atazanavir
Number analyzed (Participants) | 8 | 8 | 8
Hours
  Day 1 | 5.01 [3 to 12] | 5.05 [4 to 12] | 5 [5 to 6]
  Day 28 | 4.5 [0 to 12] | 5 [4 to 6.02] | 4.5 [3 to 6]

13. Secondary Outcome: Maximum Observed Plasma Concentrations (Cmax) - Part A and C
Description: Cmax was defined as the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Time Frame: Pre-dose Day 1 and Day 10
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter
Arm/Group | Part A-Group 1: BMS-955176 (5 mg) | Part A-Group 2: BMS-955176 (10 mg) | Part A-Group 3: BMS-955176 (20 mg) | Part A-Group 4: BMS-955176 (40 mg) | Part A-Group 9: BMS-955176 (80 mg) | Part A-Group 10: BMS-955176 (120 mg) | Part C-Group 8: BMS-955176 (40 mg) | Part C-Group 13: BMS-955176 (120 mg)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 7
Nanogram/milliliter
  Day 1 | 79.376 (37.6) | 201.498 (21.1) | 349.466 (23.2) | 791.317 (46.8) | 1155.448 (27.1) | 1515.389 (27.4) | 793.569 (21.2) | 1907.747 (38.9)
  Day 10 | 170.778 (20.8) | 337.379 (20.9) | 705.073 (15.4) | 1476.166 (17.2) | 2466.447 (22.1) | 2809.671 (25.5) | 1560.122 (17.4) | 3377.967 (32.8)

14. Secondary Outcome: Plasma Concentration 24 Hours Post-Dose (C24) - Part A and C
Description: C24 was defined as the plasma concentration of BMS-955176 at 24 hours post-dose.
Time Frame: 24 hours post-dose
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter
Arm/Group | Part A-Group 1: BMS-955176 (5 mg) | Part A-Group 2: BMS-955176 (10 mg) | Part A-Group 3: BMS-955176 (20 mg) | Part A-Group 4: BMS-955176 (40 mg) | Part A-Group 9: BMS-955176 (80 mg) | Part A-Group 10: BMS-955176 (120 mg) | Part C-Group 8: BMS-955176 (40 mg) | Part C-Group 13: BMS-955176 (120 mg)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 7
Nanogram/milliliter
  Day 1 | 34.946 (28.4) | 79.002 (27.2) | 154.5 (23.7) | 286.268 (15.6) | 482.349 (34.3) | 624.745 (24.6) | 339.173 (30.1) | 865.867 (41)
  Day 10 | 81.642 (23.1) | 138.775 (34.1) | 325.934 (19.4) | 713.077 (21.9) | 1150.397 (31.5) | 1288.985 (26.8) | 779.438 (24.6) | 1691.306 (29)

15. Secondary Outcome: Maximum Observed Plasma Concentrations (Cmax) - Part B
Description: as for outcome 13
Time Frame: Pre-dose Day 1 and Day 28
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter
Arm/Group | Part B-Group 5: BMS-955176 (40 mg) + Atazanavir | Part B-Group 6: BMS-955176 (40 mg) + Atazanavir + Ritonavir | Part B-Group 12: BMS-955176 (80 mg) + Atazanavir
Number analyzed (Participants) | 8 | 8 | 8
Nanogram/milliliter
  Day 1 | 695.596 (9.52) | 770.975 (28.2) | 1493.336 (24)
  Day 28 | 1667.817 (30.2) | 1852 (33.6) | 3159.181 (22.1)

16. Secondary Outcome: Plasma Concentration 24 Hours Post-Dose (C24) - Part B
Description: C24 was defined as the plasma concentration of BMS-955176 at 24 hours post-dose.
Time Frame: 24 hours post-dose
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter
Arm/Group | Part B-Group 5: BMS-955176 (40 mg) + Atazanavir | Part B-Group 6: BMS-955176 (40 mg) + Atazanavir + Ritonavir | Part B-Group 12: BMS-955176 (80 mg) + Atazanavir
Number analyzed (Participants) | 8 | 8 | 8
Nanogram/milliliter
  Day 1 | 462.312 (25) | 520.048 (27.7) | 899.364 (21.2)
  Day 28 | 1099.313 (37) | 1163.177 (30.9) | 2010.679 (19.9)

17. Secondary Outcome: Area Under The Plasma Concentration - Time Curve Over the Dosing Interval (AUC([Tau]) - Part A and C
Description: AUC(tau) was defined as the area under the plasma concentration - time curve over the dosing interval.
Time Frame: Pre-dose Day 1 and Day 10
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour/milliliter
Arm/Group | Part A-Group 1: BMS-955176 (5 mg) | Part A-Group 2: BMS-955176 (10 mg) | Part A-Group 3: BMS-955176 (20 mg) | Part A-Group 4: BMS-955176 (40 mg) | Part A-Group 9: BMS-955176 (80 mg) | Part A-Group 10: BMS-955176 (120 mg) | Part C-Group 8: BMS-955176 (40 mg) | Part C-Group 13: BMS-955176 (120 mg)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 7
Nanogram*hour/milliliter
  Day 1 | 1151.062 (32.2) | 2869.626 (21.3) | 5132.951 (21.5) | 10088.23 (23.1) | 17057.26 (29) | 21872.72 (27) | 10936.9 (29.9) | 26753.74 (35.9)
  Day 10 | 2720.237 (20.7) | 5168.553 (23.6) | 11751.82 (15.1) | 22984.83 (17.2) | 39341.11 (24.2) | 44182.4 (27) | 25556.64 (20.4) | 53972.71 (30.2)

18. Secondary Outcome: Area Under The Plasma Concentration - Time Curve Over the Dosing Interval (AUC[Tau]) - Part B
Description: AUC(tau) was defined as the area under the plasma concentration - time curve over the dosing interval.
Time Frame: Pre-dose Day 1 and Day 28
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour/milliliter
Arm/Group | Part B-Group 5: BMS-955176 (40 mg) + Atazanavir | Part B-Group 6: BMS-955176 (40 mg) + Atazanavir + Ritonavir | Part B-Group 12: BMS-955176 (80 mg) + Atazanavir
Number analyzed (Participants) | 8 | 8 | 8
Nanogram*hour/milliliter
  Day 1 | 12147.23 (15.2) | 12954.8 (26.2) | 24478.35 (22.6)
  Day 28 | 31406.32 (31.7) | 34225.08 (30.6) | 59915.72 (16.3)

19. Secondary Outcome: Accumulation Index (AI): Part A and C
Description: Accumulation index was calculated by dividing the AUC(tau) or Cmax or C24 of BMS-955176 on Day 10 by the AUC(TAU) or Cmax or C24, respectively, of BMS-955176 on Day 1.
Time Frame: Baseline and Day 10
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part A-Group 1: BMS-955176 (5 mg) | Part A-Group 2: BMS-955176 (10 mg) | Part A-Group 3: BMS-955176 (20 mg) | Part A-Group 4: BMS-955176 (40 mg) | Part A-Group 9: BMS-955176 (80 mg) | Part A-Group 10: BMS-955176 (120 mg) | Part C-Group 8: BMS-955176 (40 mg) | Part C-Group 13: BMS-955176 (120 mg)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 7
Ratio
  Cmax | 2.152 (42.9) | 1.674 (31.1) | 2.018 (39.8) | 1.856 (33.6) | 2.135 (16.6) | 1.854 (22.7) | 1.966 (17.2) | 1.771 (42.6)
  C24 | 2.336 (21.9) | 1.757 (35) | 2.11 (29.5) | 2.491 (24.9) | 2.385 (25.1) | 2.063 (19.3) | 2.298 (28.4) | 1.953 (42.1)
  AUC | 2.363 (25.9) | 1.801 (30.4) | 2.289 (39.7) | 2.278 (28.2) | 2.306 (19) | 2.02 (19.7) | 2.337 (26.1) | 2.017 (39)

20. Secondary Outcome: Apparent Total Body Clearance: Part A and C
Description: Apparent total body clearance was derived by non-compartmental methods, using a validated pharmacokinetic (PK) analysis program: KineticaTM 5.0 within eToolbox (version 2.7).
Time Frame: Baseline (Day 1) to Day 10
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliters/minute
Arm/Group | Part A-Group 1: BMS-955176 (5 mg) | Part A-Group 2: BMS-955176 (10 mg) | Part A-Group 3: BMS-955176 (20 mg) | Part A-Group 4: BMS-955176 (40 mg) | Part A-Group 9: BMS-955176 (80 mg) | Part A-Group 10: BMS-955176 (120 mg) | Part C-Group 8: BMS-955176 (40 mg) | Part C-Group 13: BMS-955176 (120 mg)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 7
Milliliters/minute | 30.635 (18.3) | 32.246 (28) | 28.364 (15.5) | 29.005 (18.8) | 33.892 (23.8) | 45.267 (34) | 26.086 (21.3) | 37.056 (33.7)

21. Secondary Outcome: Degree of Fluctuation (DF): Part A and C
Description: DF was calculated as the difference between Cmax and Cmin divided by Css-avg. DF was derived by non-compartmental methods, using a validated pharmacokinetic (PK) analysis program: KineticaTM 5.0 within eToolbox (version 2.7).
Time Frame: Baseline (Day 1) to Day 10
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part A-Group 1: BMS-955176 (5 mg) | Part A-Group 2: BMS-955176 (10 mg) | Part A-Group 3: BMS-955176 (20 mg) | Part A-Group 4: BMS-955176 (40 mg) | Part A-Group 9: BMS-955176 (80 mg) | Part A-Group 10: BMS-955176 (120 mg) | Part C-Group 8: BMS-955176 (40 mg) | Part C-Group 13: BMS-955176 (120 mg)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 7
Ratio | 0.766 (29.4) | 0.912 (15.2) | 0.758 (20.2) | 0.78 (22.1) | 0.779 (28.5) | 0.818 (17.1) | 0.723 (13.7) | 0.727 (24.5)

22. Secondary Outcome: Average Observed Plasma Concentration at Steady State (Css-avg): Part A and C
Description: Css-avg was calculated by the quotient of AUC(TAU) and the dosing interval (24 h). Css-avg was derived by non-compartmental methods, using a validated pharmacokinetic (PK) analysis program: KineticaTM 5.0 within eToolbox (version 2.7).
Time Frame: Baseline (Day 1) to Day 10
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter
Arm/Group | Part A-Group 1: BMS-955176 (5 mg) | Part A-Group 2: BMS-955176 (10 mg) | Part A-Group 3: BMS-955176 (20 mg) | Part A-Group 4: BMS-955176 (40 mg) | Part A-Group 9: BMS-955176 (80 mg) | Part A-Group 10: BMS-955176 (120 mg) | Part C-Group 8: BMS-955176 (40 mg) | Part C-Group 13: BMS-955176 (120 mg)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 7
Nanogram/milliliter | 113.326 (20.7) | 215.111 (23.8) | 489.507 (15.1) | 956.222 (17.3) | 1639.471 (24.2) | 1841.413 (27) | 1065.435 (19.9) | 2256.793 (30.2)

23. Secondary Outcome: Plasma Half-life: Part A and C
Description: Half-life of the terminal log-linear phase, (T-half), was calculated as natural logarithm of 2 (ln2)/λ, where λ is the absolute value of the slope of the terminal log-linear phase. T-half was derived by non-compartmental methods, using a validated pharmacokinetic (PK) analysis program: KineticaTM 5.0 within eToolbox (version 2.7).
Time Frame: Baseline (Day 1) to Day 10
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A-Group 1: BMS-955176 (5 mg) | Part A-Group 2: BMS-955176 (10 mg) | Part A-Group 3: BMS-955176 (20 mg) | Part A-Group 4: BMS-955176 (40 mg) | Part A-Group 9: BMS-955176 (80 mg) | Part A-Group 10: BMS-955176 (120 mg) | Part C-Group 8: BMS-955176 (40 mg) | Part C-Group 13: BMS-955176 (120 mg)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 7
Hours | 32.134 [25.45 to 46.45] | 31.967 [23.97 to 43.02] | 27.382 [24 to 41.59] | 33.475 [25.79 to 42.39] | 29.171 [24.32 to 38.02] | 34.574 [29.01 to 39.69] | 31.565 [24.39 to 51.64] | 35.278 [26.65 to 38.71]

24. Secondary Outcome: Number of Participants With Clinically Significant Grade 3/4 Laboratory Abnormalities From Baseline
Description: Laboratory abnormalities were determined and graded using the Division of Acquired Immune Deficiency Syndrome (AIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, version 1.0, December 2004.
Time Frame: Day 1 to up to end of the study (Day 42)
Population: All Treated Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-Group 1: BMS-955176 (5 mg) | Part A-Group 2: BMS-955176 (10 mg) | Part A-Group 3: BMS-955176 (20 mg) | Part A-Group 4: BMS-955176 (40 mg) | Part A-Group 9: BMS-955176 (80 mg) | Part A-Group 10: BMS-955176 (120 mg) | Part B-Group 5: BMS-955176 (40 mg) + Atazanavir | Part B-Group 6: BMS-955176 (40 mg) + Atazanavir + Ritonavir | Part B-Group 7: Atazanavir+Ritonavir+Tenofovir+Emtricitabine | Part B-Group 12: BMS-955176 (80 mg) + Atazanavir | Part C-Group 8: BMS-955176 (40 mg) | Part C-Group 13: BMS-955176 (120 mg) | Placebo Clade B | Placebo Clade C
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 4 | 8 | 8 | 7 | 12 | 4
Participants
  Neutrophils (Absolute) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Bilirubin (Total) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 5 | 3 | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Number of Participants With Clinically Significant Changes in Heart Rate
Description: Heart rate was measured after the participants had been seated quietly for at least 5 minutes. Criteria used to determine heart rate that are outside of a pre-specified range, where changes from Baseline are based on matched postural positions and are calculated as parameter value - Baseline parameter value: Value >100 and change from Baseline > 30, or Value < 55 and change from Baseline < -15.
Time Frame: Day 1 to end of the study (Day 42)
Population: All Treated Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-Group 1: BMS-955176 (5 mg) | Part A-Group 2: BMS-955176 (10 mg) | Part A-Group 3: BMS-955176 (20 mg) | Part A-Group 4: BMS-955176 (40 mg) | Part A-Group 9: BMS-955176 (80 mg) | Part A-Group 10: BMS-955176 (120 mg) | Part B-Group 5: BMS-955176 (40 mg) + Atazanavir | Part B-Group 6: BMS-955176 (40 mg) + Atazanavir + Ritonavir | Part B-Group 7: Atazanavir+Ritonavir+Tenofovir+Emtricitabine | Part B-Group 12: BMS-955176 (80 mg) + Atazanavir | Part C-Group 8: BMS-955176 (40 mg) | Part C-Group 13: BMS-955176 (120 mg) | Placebo Clade B | Placebo Clade C
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 4 | 8 | 8 | 7 | 12 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0

26. Secondary Outcome: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG)
Description: Participants with out of range ECG intervals were summarized. Criteria used to determine ECG results that are outside of a pre-specified range: PR (milliseconds [msec]): Value >200; QRS (msec): Value >120; QT (msec): Value >500 or change from Baseline >30; corrected QT interval Fridericia's formula (QTcF) (msec): Value >450 or change from Baseline >30.
Time Frame: Day 1 to end of the study (Day 42)
Population: All Treated Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-Group 1: BMS-955176 (5 mg) | Part A-Group 2: BMS-955176 (10 mg) | Part A-Group 3: BMS-955176 (20 mg) | Part A-Group 4: BMS-955176 (40 mg) | Part A-Group 9: BMS-955176 (80 mg) | Part A-Group 10: BMS-955176 (120 mg) | Part B-Group 5: BMS-955176 (40 mg) + Atazanavir | Part B-Group 6: BMS-955176 (40 mg) + Atazanavir + Ritonavir | Part B-Group 7: Atazanavir+Ritonavir+Tenofovir+Emtricitabine | Part B-Group 12: BMS-955176 (80 mg) + Atazanavir | Part C-Group 8: BMS-955176 (40 mg) | Part C-Group 13: BMS-955176 (120 mg) | Placebo Clade B | Placebo Clade C
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 4 | 8 | 8 | 7 | 12 | 4
Participants
  PR > 200 msec | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0
  QRS > 120 msec | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QT > 500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcB > 450 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  QTcF > 450 msec | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

27. Secondary Outcome: Number of Participants With Abnormal Changes in Physical Examination
Description: Participants with abnormal changes in physical examination is presented.
Time Frame: Day 1 to end of the study (Day 42)
Population: All Treated Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-Group 1: BMS-955176 (5 mg) | Part A-Group 2: BMS-955176 (10 mg) | Part A-Group 3: BMS-955176 (20 mg) | Part A-Group 4: BMS-955176 (40 mg) | Part A-Group 9: BMS-955176 (80 mg) | Part A-Group 10: BMS-955176 (120 mg) | Part B-Group 5: BMS-955176 (40 mg) + Atazanavir | Part B-Group 6: BMS-955176 (40 mg) + Atazanavir + Ritonavir | Part B-Group 7: Atazanavir+Ritonavir+Tenofovir+Emtricitabine | Part B-Group 12: BMS-955176 (80 mg) + Atazanavir | Part C-Group 8: BMS-955176 (40 mg) | Part C-Group 13: BMS-955176 (120 mg) | Placebo Clade B | Placebo Clade C
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 4 | 8 | 8 | 7 | 12 | 4
Participants
  Height | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Weight | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Body mass index | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

28. Secondary Outcome: Number of Participants With Clinically Significant Changes in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Systolic BP (millimeter of mercury [mmHg]): value >140 and change from Baseline >20, or value <90 and change from Baseline <-20; Diastolic BP (mmHg): value >90 and change from Baseline >10, or value <55 and change from Baseline <-10.
Time Frame: Day 1 to end of the study (Day 42)
Population: All Treated Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-Group 1: BMS-955176 (5 mg) | Part A-Group 2: BMS-955176 (10 mg) | Part A-Group 3: BMS-955176 (20 mg) | Part A-Group 4: BMS-955176 (40 mg) | Part A-Group 9: BMS-955176 (80 mg) | Part A-Group 10: BMS-955176 (120 mg) | Part B-Group 5: BMS-955176 (40 mg) + Atazanavir | Part B-Group 6: BMS-955176 (40 mg) + Atazanavir + Ritonavir | Part B-Group 7: Atazanavir+Ritonavir+Tenofovir+Emtricitabine | Part B-Group 12: BMS-955176 (80 mg) + Atazanavir | Part C-Group 8: BMS-955176 (40 mg) | Part C-Group 13: BMS-955176 (120 mg) | Placebo Clade B | Placebo Clade C
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 4 | 8 | 8 | 7 | 12 | 4
Participants
  SBP | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  DBP | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Day 1 to up to end of the study (Day 42)
Description: All Treated Subjects comprised of all participants who had received at least one dose of study medication were analyzed.
Arm/Group | Part A-Group 1: BMS-955176 (5 mg) | Part A-Group 2: BMS-955176 (10 mg) | Part A-Group 3: BMS-955176 (20 mg) | Part A-Group 4: BMS-955176 (40 mg) | Part A-Group 9: BMS-955176 (80 mg) | Part A-Group 10: BMS-955176 (120 mg) | Placebo Clade B | Part B-Group 5: BMS-955176 (40 mg) + Atazanavir | Part B-Group 6: BMS-955176 (40 mg) + Atazanavir + Ritonavir | Part B-Group 7: Atazanavir+Ritonavir+Tenofovir+Emtricitabine | Part B-Group 12: BMS-955176 (80 mg) + Atazanavir | Part C-Group 8: BMS-955176 (40 mg) | Part C-Group 13: BMS-955176 (120 mg) | Placebo Clade C
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/12 | 0/8 | 0/8 | 0/4 | 0/8 | 0/8 | 0/7 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/12 | 0/8 | 0/8 | 0/4 | 0/8 | 0/8 | 0/7 | 0/4
Other Adverse Events (participants affected / at risk) | 5/8 | 5/8 | 5/8 | 6/8 | 8/8 | 7/8 | 9/12 | 8/8 | 8/8 | 4/4 | 6/8 | 7/8 | 6/7 | 3/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A-Group 1: BMS-955176 (5 mg) (N=8) | Part A-Group 2: BMS-955176 (10 mg) (N=8) | Part A-Group 3: BMS-955176 (20 mg) (N=8) | Part A-Group 4: BMS-955176 (40 mg) (N=8) | Part A-Group 9: BMS-955176 (80 mg) (N=8) | Part A-Group 10: BMS-955176 (120 mg) (N=8) | Placebo Clade B (N=12) | Part B-Group 5: BMS-955176 (40 mg) + Atazanavir (N=8) | Part B-Group 6: BMS-955176 (40 mg) + Atazanavir + Ritonavir (N=8) | Part B-Group 7: Atazanavir+Ritonavir+Tenofovir+Emtricitabine (N=4) | Part B-Group 12: BMS-955176 (80 mg) + Atazanavir (N=8) | Part C-Group 8: BMS-955176 (40 mg) (N=8) | Part C-Group 13: BMS-955176 (120 mg) (N=7) | Placebo Clade C (N=4)
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site related reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sensation of foreign body (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 3 | 1 | 3 | 3 | 3 | 3 | 3 | 0 | 3 | 2 | 0 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mood swings (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysmenorrhea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 6 | 8 | 4 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin unconjugated increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intraocular pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 3 | 0 | 5 | 4 | 5 | 5 | 5 | 3 | 2 | 4 | 4 | 2 | 3
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Poor quality sleep (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular icterus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Foreign body sensation in eyes (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
External ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 3 | 2 | 2 | 3 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faeces hard (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 3 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gonorrhoea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulpitis dental (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.